CLINICAL TRIAL: NCT03643705
Title: A Nurse-led Intervention to Extend the HIV Treatment Cascade for Cardiovascular Disease Prevention
Acronym: EXTRA-CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Duke University (Other); University Hospitals Cleveland Medical Center (Other); MetroHealth Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Chris Todd Longenecker, Associate Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03-18-16; U01HL142099 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS; Hypertension; Hyperlipidemias
Keywords: Implementation Science; Cardiovascular Disease; Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension; Hyperlipidemias; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Intervention (Experimental): This multi-component intervention will consist of four evidence-based components delivered at 4 in-person visits (0, 4, 8, and 12 months) and by telephone contact: (1) nurse-led care coordination, (2) nurse-managed medication protocols and adherence support (3) home blood pressure monitoring, and (4) electronic medical records support tools.
  Interventions: Other: Multi-component intervention
- Education Control (Active Comparator): Participants in the education control arm will receive general prevention education delivered at 4 in-person visits (0, 4, 8, and 12 months), which will consist of evidence-based material on diet, exercise, smoking, sexually transmitted infections, and cancer prevention.
  Interventions: Other: General prevention education

INTERVENTIONS:
Other: Multi-component intervention — 4 components as described
  Arms: Nurse Intervention
Other: General prevention education — General education as described
  Arms: Education Control

SUMMARY:
Strategies to improve uptake of cardiovascular disease preventive therapies among people living with HIV (PLHIV) are urgently needed. This study tests an innovative prevention nurse intervention to extend the HIV/AIDS treatment cascade for the treatment of hypertension and hyperlipidemia among PLHIV on suppressive antiretroviral therapy. This intervention may be scalable as an extension of ongoing HIV/AIDS treatment cascade initiatives in HIV specialty clinics nationwide.

DETAILED DESCRIPTION:
People living with HIV (PLHIV) are at increased risk for atherosclerotic cardiovascular disease (ASCVD); however, uptake of evidence based therapies to prevent ASCVD is sub-optimal. Reasons for under treatment may include low perceived risk, competing priorities for HIV specialist providers, and poor trust and communication with non-HIV primary care providers. This project proposes a nurse-led intervention to extend the HIV/AIDS treatment cascade-a widely adopted framework developed to improve access to high quality HIV care-for CVD prevention, specifically to improve control of blood pressure and hyperlipidemia in PLHIV on antiretroviral therapy who have suppressed HIV viral load. The study will be conducted in three racially and ethnically diverse clinic contexts [University Hospitals (Cleveland, OH), MetroHealth (Cleveland, OH) and Duke Health (Durham, NC)] that are broadly representative of HIV specialty care in the US. Using a mixed-methods clinical effectiveness trial design, this project will test the 12-month efficacy of a multi-component intervention among n=300 HIV+ adults on suppressive ART with hypertension and hyperlipidemia. Participants will be randomized 1:1 to intervention vs. education control. Control participants will receive general prevention education. The intervention will consist of four evidence-based components derived from prior studies in the general population: (1) nurse-led care coordination, (2) nurse-managed medication protocols and adherence support (3) home BP monitoring, and (4) electronic medical records (EMR) support tools. These components will be further adapted to the HIV specialty clinic context with key stakeholder input and using data from a mixed-methods study of current ASCVD preventive care practices at the three HIV clinic sites. A process evaluation of the prevention nurse intervention will be conducted, which will assess fidelity, dose, recruitment, reach, and context. Two key contextual process measures of interest will be changes in perceived ASCVD risk and changes in trust and communication between PLHIV participants and their HIV and non-HIV providers. If proven effective to reduce both blood pressure and cholesterol as postulated, this nurse-led intervention will have substantial clinical impact among high-risk PLHIV, potentially reducing ASCVD events by more than a quarter. This model is potentially scalable as an extension of HIV treatment cascade initiatives nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Laboratory confirmed HIV+ diagnosis
3. Undetectable HIV viral load: defined as the most recent HIV viral load <200 copies/mL, checked within the past year (assessed via chart abstraction)
4. Hypertension: defined as systolic blood pressure >130 mmHg on ≥ 2 occasions in the past 12 months or on an antihypertensive medication (assessed via chart abstraction)
5. Hyperlipidemia: defined as a non-high-density lipoprotein cholesterol level >130mg/dL or on cholesterol lowering medication

Exclusion Criteria:

1. On lipid-lowering medication solely for cardiovascular disease prevention with evidence of pre-medication non-high-density lipoprotein cholesterol which was already below 100mg/dL
2. On anti-hypertensive medications solely for a non-hypertension indication (e.g. systolic heart failure)
3. Severely hearing or speech impaired, or other disability that would limit participation in the intervention components
4. In a nursing home and/or receiving in-patient psychiatric care
5. Terminal illness with life expectancy < 4 months
6. No reliable access to a telephone
7. Pregnant, breast-feeding, or planning a pregnancy during the study period
8. Planning to move out of the area in the next 12 months
9. Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris T Longenecker, MD, Principal Investigator — University of Washington; Allison R Webel, RN PhD, Principal Investigator — University of Washington; Hayden Bosworth, PhD, Principal Investigator — Duke University; Barb Gripshover, MD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - Duke Health, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
In collaboration with the National Institutes of Health funding body, we will develop a process to facilitate providing other investigators with access to appropriately de-identified study data. We will make the following available upon request after the primary manuscript is published: de-identified data set, trial description information, data collection forms, and data structure.
Time Frame: After publication of the primary manuscript
Access Criteria: Data will be made available upon request or on a data share site after publication of the primary manuscript.

REFERENCES:
- [Derived] Longenecker CT, Jones KA, Hileman CO, Okeke NL, Gripshover BM, Aifah A, Bloomfield GS, Muiruri C, Smith VA, Vedanthan R, Webel AR, Bosworth HB. Nurse-Led Strategy to Improve Blood Pressure and Cholesterol Level Among People With HIV: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e2356445. doi: 10.1001/jamanetworkopen.2023.56445. PMID 38441897
- [Derived] Schexnayder J, Longenecker CT, Muiruri C, Bosworth HB, Gebhardt D, Gonzales SE, Hanson JE, Hileman CO, Okeke NL, Sico IP, Vedanthan R, Webel AR. Understanding constraints on integrated care for people with HIV and multimorbid cardiovascular conditions: an application of the Theoretical Domains Framework. Implement Sci Commun. 2021 Feb 12;2(1):17. doi: 10.1186/s43058-021-00114-z. PMID 33579396
- [Derived] Webel AR, Schexnayder J, Rentrope CR, Bosworth HB, Hileman CO, Okeke NL, Vedanthan R, Longenecker CT. The influence of healthcare financing on cardiovascular disease prevention in people living with HIV. BMC Public Health. 2020 Nov 23;20(1):1768. doi: 10.1186/s12889-020-09896-8. PMID 33228623
- [Derived] Okeke NL, Webel AR, Bosworth HB, Aifah A, Bloomfield GS, Choi EW, Gonzales S, Hale S, Hileman CO, Lopez-Kidwell V, Muiruri C, Oakes M, Schexnayder J, Smith V, Vedanthan R, Longenecker CT. Rationale and design of a nurse-led intervention to extend the HIV treatment cascade for cardiovascular disease prevention trial (EXTRA-CVD). Am Heart J. 2019 Oct;216:91-101. doi: 10.1016/j.ahj.2019.07.005. Epub 2019 Jul 18. PMID 31419622

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nurse Intervention | Education Control
Started | 149 | 148
Completed | 114 | 129
Not Completed | 35 | 19

BASELINE CHARACTERISTICS:
Population: 1 participant withdrew after randomization but before the baseline data collection occurred
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Intervention | Education Control | Total
Number analyzed (Participants) | 149 | 148 | 297
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [53 to 65] | 59.5 [52.5 to 64] | 59 [53 to 65]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 113 | 120 | 233
  Transgender Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 79 | 97 | 176
  White | 60 | 41 | 101
  Other race | 4 | 5 | 9
  Multiracial | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 148 | 297
Number of Participants Enrolled at Each Site [Count of Participants; unit: Participants] — Site reporting is anonymous (i.e. Site A, B, and C) as per IRB protocol to protect the participating sites
  Participants
    Site A | 49 | 50 | 99
    Site B | 50 | 50 | 100
    Site C | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Repeated measures across 4 time points (0, 4, 8, and 12 months)
Time Frame: 12 months
Measure: Mean (Standard Error); unit: model estimated mmhg
Arm/Group | Nurse Intervention | Education Control
Number analyzed (Participants) | 149 | 148
model estimated mmhg
  Baseline | 134.9 (1.0) | 134.9 (1.0)
  4 months | 129.9 (1.5) | 136.3 (1.5)
  8 months | 129.3 (1.6) | 133.0 (1.4)
  12 months | 129.7 (1.5) | 133.9 (1.4)

2. Secondary Outcome: Non High Density Lipoprotein (Non-HDL) Cholesterol
Description: Repeated measures across 4 time points (0, 4, 8, and 12 months)
Time Frame: 12 months
Measure: Mean (Standard Error); unit: model estimated mg/dL
Arm/Group | Nurse Intervention | Education Control
Number analyzed (Participants) | 149 | 148
model estimated mg/dL
  Baseline | 139.9 (2.5) | 139.9 (2.5)
  4 months | 127.4 (3.5) | 135.7 (3.4)
  8 months | 120.9 (3.5) | 131.9 (3.3)
  12 months | 114.7 (3.5) | 132.1 (3.3)

3. Other Pre Specified Outcome: % of Subjects in Each Hypertension Cascade Category
Description: Ordinal 3-level variable across 4 time points (0, 4, 8, and 12 months). The hypertension cascade tool is reported as mutually exclusive categories as follows: 1=untreated hypertension; 2=hypertension treated; 3=blood pressure target achieved. NOTE: This differs from our protocol specified 4-level variable because the numbers in the first two categories were too small. Therefore, undiagnosed and diagnosed were collapsed into one "untreated" category.
Time Frame: 12 months
Measure: Number; unit: model estimated %
Arm/Group | Nurse Intervention | Education Control
Number analyzed (Participants) | 149 | 148
model estimated %
  Untreated Baseline | 10.8 | 10.8
  Treated Baseline | 47.3 | 47.3
  At treatment goal Baseline | 42.0 | 42.0
  Untreated 4 months | 7.8 | 9.9
  Treated 4 months | 34.3 | 45.7
  At treatment goal 4 months | 57.9 | 44.4
  Untreated 8 months | 3.2 | 7.7
  Treated 8 months | 33.2 | 45.3
  At treatment goal 8 months | 63.6 | 47.0
  Untreated 12 months | 5.7 | 11.6
  Treated 12 months | 34.4 | 48.6
  At treatment goal 12 months | 59.9 | 39.8

4. Other Pre Specified Outcome: % of Subjects in Each Hyperlipidemia Cascade Category
Description: Ordinal 3-level variable across 4 time points (0, 4, 8, and 12 months). The cholesterol cascade is reported as mutually exclusive categories as follows: 1=untreated hyperlipidemia; 2=hyperlipidemia treated; 3=non-HDL cholesterol target achieved. NOTE: This differs from our protocol specified 4-level variable because the numbers in the first two categories were too small. Therefore, undiagnosed and diagnosed were collapsed into one "untreated" category.
Time Frame: 12 months
Measure: Number; unit: model estimated %
Arm/Group | Nurse Intervention | Education Control
Number analyzed (Participants) | 149 | 148
model estimated %
  Untreated Baseline | 37.5 | 37.5
  Treated Baseline | 20.5 | 20.5
  At treatment goal Baseline | 42.0 | 42.0
  Untreated 4 months | 18.1 | 27.5
  Treated 4 months | 15.7 | 18.0
  At treatment goal 4 months | 66.3 | 54.5
  Untreated 8 months | 5.9 | 16.3
  Treated 8 months | 9.0 | 16.3
  At treatment goal 8 months | 85.1 | 67.4
  Untreated 12 months | 5.3 | 27.1
  Treated 12 months | 3.6 | 14.1
  At treatment goal 12 months | 91.1 | 58.7

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participants were assessed for adverse events systematically by the study nurse at each 4-month study visit. This included any self-reported events as well as a review of the electronic health record.
Arm/Group | Nurse Intervention | Education Control
All-Cause Mortality (participants affected / at risk) | 2/149 | 2/148
Serious Adverse Events (participants affected / at risk) | 30/149 | 22/148
Other Adverse Events (participants affected / at risk) | 44/149 | 45/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse Intervention (N=149) | Education Control (N=148)
Non-study related events (General disorders) | 26 (43) | 22 (47) — No serious adverse events were deemed to be possibly, probably, or definitely study related. Non-study related adverse events were monitored/assessed without regard to the specific Adverse Event Term
Emergency room visit or hospitalization for high home blood pressure (Vascular disorders) | 3 (3) | 0 (0)
Emergency room visit for chest pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse Intervention (N=149) | Education Control (N=148)
Acute kidney injury due to antihypertensive medication (Renal and urinary disorders) | 1 (1) | 0 (0)
myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
possible angioedema (Immune system disorders) | 1 (1) | 0 (0)
non study related events (General disorders) | 41 (41) | 45 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT03643705/Prot_SAP_000.pdf